CLINICAL TRIAL: NCT00639535
Title: Comparative Study of the Diagnostic Accuracy of Scintimammography (Fluorine 18-FDG PET Scintigraphic Imaging) and Magnetic Resonance Imaging in Identifying Malignant Breast Lesions, In Subjects With Breast Abnormalities
Brief Title: Study Comparing the PET Scan and MRI in Identifying Breast Malignancies in Women With Breast Abnormalities
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, David Feiglin, Chairman Radiology Department, State University of New York - Upstate Medical University
Other Study IDs: SUNYUMU 4493
Record Dates: First submitted 2008-03-12; First posted 2008-03-20 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Breast Disease
Keywords: Radiology; MRI; Positron emission tomography; Breast Abnormalities; Dense Breast Tissue
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study looking at advanced imaging such as PET/CT and MRI to see if they can provide a more accurate assessment of the patient with dense breasts or difficult to interpret mammograms. In addition, the ability to determine whether one or the other is more accurate or whether both together would be appropriate in this clinical situation, may be able to be measured.

The MRI studies are very sensitive for detection of breast histopathology but less specific in differentiating between small low grade malignancies are more benign pathologies. Multifocal pathology can be challenging in determining site(s) for biopsy.

PET scanning is specific in the measurement of metabolic glucose activity of various histopathologies and is accurate in differentiating aggressive from benign pathology in multifocal breast disease. A further drawback of PET is the lack of ability to observe lesions less than 3-4mm in diameter.

In select cases the combination of MR and PET/CT is able to come to a more conclusive diagnosis - specifically with bilateral or multifocal breast disease.

ELIGIBILITY:
Inclusion Criteria:

* Woman who have breast volumes allowing utilization of MRI breast coil
* Patients who are considered, by radiologist reading the mammograms, to have non interpretable or difficult to interpret x-ray studies. These patients may or may not have palpable breast lumps and may and may not have suspicious areas on their x-ray mammograms.

Exclusion Criteria:

* Women of child bearing potential not practicing a medically accepted method of birth control
* Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from Breast Care Clinic and local physicians.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2002-01 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Feiglin, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (3):
- United States (3):
  - Central New York PET Center, Liverpool, New York
  - University Radiology Associates, Syracuse, New York
  - Institute For Human Performance, Syracuse, New York